CLINICAL TRIAL: NCT04327466
Title: Effect of High Frequency Oscillatory Highflow Nasal Cannula on Desaturations and Bradycardia in Preterm Infants: A Randomized Crossover Trial
Brief Title: Effect of High Frequency Oscillatory Highflow Nasal Cannula on Desaturations and Bradycardia in Preterm Infants
Acronym: Osciflow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Osciflow
Record Dates: First submitted 2020-03-12; First posted 2020-03-31 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Apnea of Prematurity; Infant, Premature, Diseases
Keywords: Non-invasive respiratory support; Non-invasive high frequency oscillatory ventilation; Highflow nasal cannula
MeSH Terms: conditions — Apnea; Infant, Premature, Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osciflow (Experimental): Crossover sequence of experimental treatment and active comparator.
  Interventions: Device: Osciflow
- Highflow (Active Comparator): Crossover sequence of experimental treatment and active comparator.
  Interventions: Device: Highflow

INTERVENTIONS:
Device: Osciflow — Osciflow is a non-invasive high frequency oscillatory ventilation support delivered via a highflow nasal cannula for four hours (one hour wash-out, three hours measurement period).
  Arms: Osciflow
Device: Highflow — Standard highflow therapy without oscillations delivered via a highflow nasal cannula for four hours (one hour wash-out, three hours measurement period).
  Arms: Highflow

SUMMARY:
This study evaluates the effect of non-invasive high frequency oscillations applied via a highflow nasal cannula ('Osciflow') compared to highflow nasal cannula without oscillations (HF) on desaturations and bradycardia in premature infants. It uses a crossover design. Infants are randomized to begin the study with either Osciflow or HF. Both modes are applied for 4 hours. Infants are monitored with an oximetry sensor to measure peripheral oxygen saturation (SpO2) and pulse rate, and with a transcutaneous CO2-transducer. Further measurements include respiratory rate and 'Bernese pain scale' evaluated by nursing staff and Electrical Impedance Tomography (EIT) in a subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born with a gestational age of <35 weeks
* >72 hours old
* On nCPAP with PEEP 5 mbar and FiO2 <0.3

Exclusion Criteria:

* Severe congenital malformations adversely affecting life expectancy

Min Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Paired difference in the total number of desaturations and bradycardia between Osciflow and HF | 180-minute recording periods for each therapy

SECONDARY OUTCOMES:
Paired difference in respiratory rate | 180-minute recording periods for each therapy
Paired difference in heart rate | 180-minute recording periods for each therapy
Paired difference in fraction of inspired oxygen [FiO2] | 180-minute recording periods for each therapy
Paired difference in peripheral oxygen saturation [SpO2] | 180-minute recording periods for each therapy
Paired difference in the proportion of time spent with oxygen saturations < 80% | 180-minute recording periods for each therapy
Paired difference in the proportion of time spent with heart rates < 80 bpm | 180-minute recording periods for each therapy
Paired difference in the number of apneas requiring stimulation | 180-minute recording periods for each therapy
Paired difference in transcutaneous CO2 measurements | 180-minute recording periods for each therapy
Paired difference in pain assessment using 'Bernese pain scale' | 180-minute recording periods for each therapy
  Bernese Pain-Scale for Neonates (BPSN): a 9-item multidimensional pain assessment tool that includes behavioral and physiological indicators. The instrument consists of seven subjective (alertness, crying, consolation, skin color, facial expression, posture, and changes in respiratory rate) and two physiological (i.e. objective) (changes in heart rate and oxygen saturation) indicators. Each item is rated on a four point Likert scale (0, 1, 2, and 3). Higher scores indicate greater pain-related distress, and a total score of 11 or higher is considered to indicate pain.
Paired difference in end-expiratory lung impedance (EELI) in a subset of patients. | At the end of each intervention period
  EELI using electrical impedance tomography (arbitrary units per kilogram).
Paired difference in regional ventilation distribution in a subset of patients. | At the end of each intervention period
  Regional ventilation distribution using electrical impedance tomography (arbitrary units per kilogram).
Paired difference in Tidal volumes in a subset of patients. | At the end of each intervention period
  Tidal volumes using electrical impedance tomography (arbitrary units per kilogram).
Paired difference in nasal trauma score | At the end of each intervention period
  Royal Women's Hospital Nasal Integrity and Pressure Chart.
  Nasal injury is defined as stage 0-skin intact; stage 1-nonblanchable erythema of intact skin; stage 2-partial thickness skin loss involving epidermis, dermis, or both; stage 3-full thickness skin loss involving damage to or necrosis of subcutaneous tissue; stage 4-full thickness skin loss with extensive destruction, tissue necrosis, or damage to supporting structures.
  Lowest Score: 0. Highest Score: 4. A higher score indicates more extensive nasal injury.
Paired difference in the rate of pneumothorax | 180-minute recording periods for each therapy
Paired difference in reaching 'failure criteria' to stop Osciflow or HF therapy: | 180-minute recording periods for each therapy
  Definition of failure criteria
  * Respiratory rate >90/min for more than 30 minutes
  * Respiratory rate >20/min higher than at the beginning of the study
  * Increase in FiO2 by ≥ 0.25 from baseline for more than 30 minutes
  * Apnea-Score of more than 20/4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neonatology, University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rub DM, Sivieri EM, Abbasi S, Eichenwald E. Effect of high-frequency oscillation on pressure delivered by high flow nasal cannula in a premature infant lung model. Pediatr Pulmonol. 2019 Nov;54(11):1860-1865. doi: 10.1002/ppul.24459. Epub 2019 Jul 24. PMID 31339005
- [Background] Sivieri EM, Eichenwald E, Bakri SM, Abbasi S. Effect of high frequency oscillatory high flow nasal cannula on carbon dioxide clearance in a premature infant lung model: A bench study. Pediatr Pulmonol. 2019 Apr;54(4):436-443. doi: 10.1002/ppul.24216. Epub 2018 Dec 14. PMID 30549451